CLINICAL TRIAL: NCT07120620
Title: PriCoTTF Study: A Phase I/II Study With TTFields Before and During Radiotherapy in Newly Diagnosed Glioblastoma
Brief Title: PriCoTTF Study: TTFields Before and During Radiotherapy for Newly Diagnosed Glioblastoma
Acronym: PriCoTTF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sied Kebir (Other)
Responsible Party: Sponsor-Investigator, Sied Kebir, PD. Dr. med., Head of Clinical Neuro-Oncology, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXT-201701
Record Dates: First submitted 2025-06-16; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma Multiforme (GBM)
Keywords: newly-diagnosed glioblastoma; TTFields; Tumor Treating Fields; radiotherapy; chemotherapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: surgery, TTFields, radiotherapy and chemotherapy (Experimental): Following diagnosis of primary glioblastoma, patients are treated with postsurgical TTFields (2-4 weeks after surgery and 1-2 weeks prior radiotherapy) followed by TTFields concomitant to radiotherapy (60 Gy will be given in 30 fractions with 2 Gy per fraction). Concomitant and adjuvant chemotherapy will be administered according to institutional standards and interdisciplinary tumor conference.
  Interventions: Device: TTFields before and during radiotherapy
- Arm B: Surgery, TTFields, hypofractional radiotherapy, chemotherapy (if applicable) (Experimental): Following diagnosis of primary glioblastoma, patients are treated with postsurgical TTFields (2-4 weeks after surgery and 1-2 weeks prior radiotherapy) followed by TTFields concomitant to radiotherapy for 3 weeks (40 Gy will be given at 2,67 Gy per daily fraction). Chemotherapy will be administered according to institutional standards and interdisciplinary tumor conference.
  Interventions: Device: TTFields before and during radiotherapy

INTERVENTIONS:
Device: TTFields before and during radiotherapy — Administration of TTFields before and during radiation therapy in patients with primary glioblastoma (Arm A)
  Arms: Arm A: surgery, TTFields, radiotherapy and chemotherapy
Device: TTFields before and during radiotherapy — Administration of TTFields before and during radiation therapy in patients with primary glioblastoma (Arm B)
  Arms: Arm B: Surgery, TTFields, hypofractional radiotherapy, chemotherapy (if applicable)

SUMMARY:
The PriCoTTF clinical trial is related to the development and validation of the investigational product Optune®, a device for generating tumor therapy fields (TTFields) that is used in combination with radiation therapy to treat newly diagnosed glioblastoma. The trial aims to evaluate the safety of early and concurrent use of TTFields with standard radiation chemotherapy. This strategy is based on preclinical data suggesting that TTFields increase the sensitivity of tumor cells to radiation therapy. Critical components of this clinical trial include demonstrating the safety and tolerability of TTFields in combination with radiation therapy and collecting initial efficacy data. The target population consists of patients with newly diagnosed glioblastoma, with treatment beginning immediately after surgical resection and continuing for up to nine months. Follow-up examinations will be conducted at regular intervals to monitor long-term treatment success. The trial protocol was developed in accordance with the guidelines of the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP). In addition, discussions were held between the sponsor, Essen University Hospital, and the relevant regulatory authorities to ensure that the clinical trial complies with regulatory requirements and is ethically acceptable. Compliance with these standards ensures scientific validity and patient safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Pathological evidence of glioblastoma or gliosarcoma using latest World Health Organization (WHO) classification criteria
* Negative isocitrate dehydrogenase (IDH) status on immunohistochemistry or sequencing
* Patient received brain tumor resection or biopsy and further treatment regime foresees radiotherapy with or without concomitant chemotherapy
* General indication for whole treatment regimen was a common decision of a multidisciplinary team within brain tumor board and in accordance with the national and/or international guidelines for the treatment of glioblastoma patients
* KPS ≥ 60% (Study arm A), KPS ≥ 50% (Study arm B)
* Life expectancy at least 3 months
* Participants of child-bearing age must use effective contraception
* Treatment with Tumor Treating Fields (TTFields) may start 2-4 weeks post resection and 1-2 weeks prior to radiotherapy
* Subjects with the ability to follow study instructions and likely to attend and complete all required visits
* Written informed consent of the subject

Exclusion Criteria:

General Exclusion Criteria:

* Subjects not able to give consent
* Subject without legal capacity who is unable to understand the nature, scope, significance, and consequences of this clinical trial
* Simultaneously participation in another clinical trial or participation in any clinical trial involving administration of an investigational medicinal product within 30 days prior to clinical trial beginning
* Subjects with a physical or psychiatric condition which at the investigator´s discretion may put the subject at risk, may confound the trial results or may interfere with the subject's participation in this clinical trial
* Known or persistent abuse of medication, drugs or alcohol

Exclusion criteria regarding special restrictions for females:

* Current or planned pregnancy or nursing women
* Females of child-bearing potential, who are not using and not willing to use medically reliable methods of contraception for the entire study duration (such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized / hysterectomized or there are any other criteria considered sufficiently reliable by the investigator in individual cases

Indication-specific exclusion criteria:

* Infra-tentorial tumor
* Significant comorbidities at baseline, which would prevent possible chemotherapy, including:

  * Platelet count < 100/nl
  * Absolute neutrophil count (ANC) < 1.5/nl
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal
  * Total bilirubin above the normal range
  * Serum creatinine > 1.7 mg/dl
* Patients with clinically significant liver-, renal- or blood disorder
* Patients with known additional significant neurological disease (e.g. primary seizure disorder*, dementia, progressive degenerative neurological disease, meningitis or encephalitis, hydrocephalus with increased intracranial pressure)

  *Patients with brain tumor-related epilepsy, seizure-free under antiepileptic therapy are eligible
* Documented allergy to conductive hydrogel (e.g. ECG (electrocardiogram) sticker or TENS (transcutaneous electrical nerve stimulation) electrodes
* Active implanted medical device (e.g. deep brain stimulators, spinal cord stimulators, vagus nerve stimulators, pacemakers, defibrillators and programmable shunts)or documented clinically significant arrhythmias
* Skull defect (e.g. missing bone with no replacement) and bullet fragments in the skull
* History of hypersensitivity reaction to temozolomide or lomustine
* Positive human immunodeficiency virus (HIV) Test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety (frequency of predefined treatment-limiting toxicities (TLTs)) of Tumor Treating Fields (TTFields) before and concurrently with radiation therapy in patients with primary glioblastoma | From the day of surgery until 4 weeks after end of radiotherapy (usually 10-12 weeks)
  The primary endpoint is safety and tolerability. It is based on the frequency of predefined treatment-limiting toxicities (TLTs), which are assessed weekly during therapy and up to four weeks after the end of radiation therapy.

SECONDARY OUTCOMES:
Long-term treatment-limiting toxicities (TLTs) | Until the end of treatment or tumor recurrence, whichever occurs first (usually 6 to 24 months)
  TLT 4 weeks after radiotherapy completion until the end of treatment or tumor recurrence, whichever occurs first (overall and considering concomitant chemotherapy)
Short-term treatment-limiting toxicities (TLTs) | During (usually 3-6 weeks) radiotherapy and up to 4 weeks after the end of radiotherapy
  TLT during treatment and up to 4 weeks after end of radiotherapy concomitant chemotherapy
Progession free survival (PFS) | Until tumor recurrence (usually 6 to 12 months)
  Time from diagnosis to MRI based tumor progression
Overall survival (OS) | From tumor diagnosis to death (usually 6 to 24 months)
  Overall survival from diagnosis to death
Radiological response (RANO criteria) | Until the end of treatment or tumor recurrence, whichever occurs first (usually 6 to 24 months)
  The radiological response is assessed during regular MRI follow-up examinations.
Adverse events as measured by Common Terminology Criteria for Adverse Events (CTCAE) | Until the end of treatment or tumor recurrence, whichever occurs first (usually 6 to 24 months)
  Adverse events are classified according to CTCAE
Quality of life (QoL) | At end of radiotherapy (usually 3-10 weeks after randomization); 4 weeks after the end of radiotherapy; at 3, 5 and 7 months of TTFields treatment
  The following questionnaires are used to assess quality of life:
  EORTC Core Quality of Life Questionnaire [QLQ-C30], (Part A with 28 questions on a Likert scale, 28 to 112 points, Higher score means lower quality of life; Part B with 2 questions on a Likert scale, 2 to 14 points, Lower score means lower quality of life)
  EORTC Brain Questionaire [QLQ-BN20], (20 questions on a Likert scale; 20 to 80 points; Higher score means lower quality of life)
Estimation number of fully compliant patients | Usually 7 to 12 weeks
  Fully compliant is defined as: Wearing rate of TTFields must be at least 50% between randomisation and visit 4 (4 weeks after the end of radiotherapy).
Estimation of the delivered cumulative dose distribution | From beginning to the end of radiotherapy (usually 3-6 weeks)
  Estimation of the delivered cumulative dose distribution over the treatment series for each patient from the KV-image guidance data and comparison with the planned dose distribution. Dose deviations by more than 3.5% in more than 1 cm3 within the PTV or if more than 5% in less than 1 cm3 will be considered as relevant
Number of patients with ≥ grade 3 skin toxicity (Common Terminology Criteria for Adverse Events, CTCAE) | Until the end of treatment or tumor recurrence, whichever occurs first (usually 6 to 24 months)
  Number of patients with ≥ grade 3 skin toxicity (CTCAE) separately into patients with high 1 and low radiation risk. 1: high risk group: patients who received a surface dose >70% of the prescribed dose within or up to 6 mm below the skin on a scalp area are of >50 cm2

OTHER OUTCOMES:
Exploratory endpoint: Frequency of grade 1-4 white matter lesions | at 4 weeks (Visit 4) and 6 months (Visit 7) or tumor progression (Visit P) after the end of radiotherapy (usually 6 to 12 months)
  Frequency of grade 1-4 white matter lesions at 4 weeks (Visit 4) and 6 months (Visit 7) or tumor progression (Visit P) after the end of radiotherapy until tumor progression (MRI according to visit schedule)
Exploratory endpoint: Assessment of Tumor Progression Patterns | At progression (usually 6 to 12 months)
  An investigation of tumor progression patterns will be conducted with regard to specific characteristics under experimental therapy.
Exploratory endpoint: Progression free survival (PFS) from first to second tumor progression | First to second progression (usually after 6 to 24 monts)
  PFS from first to second tumor progression (under consideration of TTFields re-challenge)
Exploratory endpoint: Overall survival (OS) | First to second progression (usually 6 to 24 monts)
  OS from first to second tumor progression (under consideration of TTFields re-challenge)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Department of Neurology, Division of Clinical Neuro-Oncology, Essen, Northrhine-Westfalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR